CLINICAL TRIAL: NCT03383848
Title: Evaluation of Patient Experience and Quality of Life During In Vitro Fertilization Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Michael Lanham, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM00121481
Record Dates: First submitted 2017-12-19; First posted 2017-12-26 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Software Group (Experimental): Subjects in the experimental group will be provided with free access to the medication management software online, which will be able to be accessed on the SmartPhone/SmartDevice and home tablet(s) or computer(s) of their choice, through any browser. They will also be provided with links to the surveys to be filled out in the REDCap secure web application throughout the study.
  Interventions: Device: Medication Management Software
- Control Group (No Intervention): Subjects in the control group will receive standard of care, and will receive emails with links to the surveys to be filled out in the REDCap secure web application throughout the study.

INTERVENTIONS:
Device: Medication Management Software — The OnTrack Medication Management Software allows patients to track the amount of fertility medication they have at home. When they check off their "to do" list of medications, it decrements the amount they have at home. It allows them to see when they will run out of medication depending on their current doses (which can change daily). Daily use of the software will be 5-10 minutes daily for approximately 21 days.
  Arms: Experimental Software Group

SUMMARY:
This study will evaluate if an electronic medication management software solution can improve outcomes for patients undergoing in vitro fertilization (IVF) treatment. Participants will be randomized equally into two groups: half will use the management software, while the other half will act as a control group.

DETAILED DESCRIPTION:
In the United States, individuals suffering from infertility pursued approximately 190,000 cycles of in vitro fertilization (IVF) in 2014, with approximately 1.5 million cycles performed internationally. Without insurance coverage, each cycle can cost between $15,000 and $25,000 for medications and procedures. The goal of an IVF cycle is a healthy baby, but to achieve this goal, patients and their partners are asked to manage administration and inventory of between 6 and 12 medications with doses and routes that can change daily. Due to the complexity of the treatment and the fact that the medications are expensive and ordered by patients incrementally to reduce large amounts of waste, medication errors (wrong dose; missed dose; running out of medication) are common (3-15% of patients).

The current standard is that patients manage this process of medication inventory, administration, and refills on their own with their own systems, using paper calendars provided by a clinic (which are immediately inaccurate once the cycle starts), paper-and-pencil lists, electronic lists, or generic medication-tracking applications, combined with verbal and written reminders from their clinic. Not having the right medication at the right time is the most critical error, and with the current methods, the patient often does not realize this fact while there is sufficient time to rectify the inventory problem, and the clinic has no way to catch at-risk patients proactively. For these patients, this error can mean a sub-optimal response with a lower chance of pregnancy that particular month (as low as 0%, depending on the error). Of the patients undergoing IVF with perfect adherence, only about 50% achieve the goal of a healthy baby. For the remainder, there will always be the concern that perhaps they could have had a different outcome, and for those with a medication error, they will never know whether the outcome could have been different if that error had not occurred.

This study will determine if patients using medication management software will have lower numbers of documented medication errors (as captured through the software and/or reported by the patient to the clinical team caring for them during their IVF cycle) compared to patients who use standard paper/pencil or home-grown methods to track their medication inventory.

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing IVF cycle (planning egg retrieval) at University of Michigan, for any indication (infertility, fertility preservation, or genetic disorder planning preimplantation genetic screening or diagnosis)
* English as primary language
* Owns a smartphone
* Owns a non-smartphone device with access to the internet at home (tablet, laptop computer, or desktop computer)
* Has internet access at home

Exclusion Criteria:

* Non-English speaker as primary language
* Previous participant in same study
* Not undergoing IVF fertility treatment
* Does not own a smartphone
* Does not own a tablet, laptop computer, or desktop computer
* Does not have internet access at home

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Documented Medication Errors | End of treatment cycle, between day 9 and day 15
  Common medication errors such as wrong dose, missed dose, or running out of medication, as captured through the software and/or reported by the patient to the clinical team caring for them during their IVF cycle.

SECONDARY OUTCOMES:
Number of Phone and Patient Portal Messages to Infertility Nurses | End of treatment cycle, between day 9 and day 15
  Number of phone and patient portal (electronic health record) messages to infertility nurses from patients using the software as compared to those using standard pencil/paper or homegrown methods to track medication inventory.
Quantity of Medication Waste | End of treatment cycle, between day 9 and day 15
  Amount of medication patient has left at the end of the IVF cycle, as an indication of medication tracking errors.
Stress Level | Baseline, between stimulation days 6 and 8, and on the day prior to egg retrieval (between day 9 and day 15 of treatment cycle)
  Change in stress levels as measured by CART (Concerns of Women Undergoing Assisted Reproductive Technologies) survey.
Anxiety Level | Baseline, between stimulation days 6 and 8, and on the day prior to egg retrieval (between day 9 and day 15 of treatment cycle)
  Change in state anxiety score as measured by Spielberger's State-Trait Anxiety Inventory survey.
Quality of Life | Baseline, between stimulation days 6 and 8, and on the day prior to egg retrieval (between day 9 and day 15 of treatment cycle)
  Change in quality of life assessment as measured by FertiQoL (Fertility Patient Quality of Life) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lanham, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Center for Reproductive Medicine, University of Michigan, Ann Arbor, Michigan
  - Northville Health Center, Northville, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin CE, Lanham M, Almgren-Bell A, Marsh C, Omurtag K. A randomized controlled trial to evaluate the use of a web-based application to manage medications during in vitro fertilization. Fertil Steril. 2021 Sep;116(3):793-800. doi: 10.1016/j.fertnstert.2021.04.022. Epub 2021 May 18. PMID 34016436